CLINICAL TRIAL: NCT01131013
Title: A Phase II, Double-Blind, Randomized, Placebo-Controlled, Three-Way Crossover, Pharmacokinetic and Pharmacodynamic Study of CK-2017357 in Patients With Claudication
Brief Title: A Study of CK-2017357 in Patients With Peripheral Artery Disease and Symptomatic Claudication
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CY 4022
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Intermittent Claudication; Peripheral Artery Disease
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease | interventions — CK-2017357

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment Sequence 1 (Experimental): Dosing Period 1 - Placebo; Dosing Period 2 - 375 mg CK-2017357; Dosing Period 3 - 500 mg CK-2017357
  Interventions: Drug: Placebo; Drug: 375 mg CK-2017357; Drug: 500 mg CK-2017357
- Treatment Sequence 2 (Experimental): Dosing Period 1 - Placebo; Dosing Period 2 - 500 mg CK-2017357; Dosing Period 3 - 375 mg CK-2017357
  Interventions: Drug: Placebo; Drug: 375 mg CK-2017357; Drug: 500 mg CK-2017357
- Treatment Sequence 3 (Experimental): Dosing Period 1 - 375 mg CK-2017357; Dosing Period 2 - Placebo; Dosing Period 3 - 500 mg CK-2017357
  Interventions: Drug: Placebo; Drug: 375 mg CK-2017357; Drug: 500 mg CK-2017357
- Treatment Sequence 4 (Experimental): Dosing Period 1 - 375 mg CK-2017357; Dosing Period 2 - 500 mg CK-2017357; Dosing Period 3 - Placebo
  Interventions: Drug: Placebo; Drug: 375 mg CK-2017357; Drug: 500 mg CK-2017357
- Treatment Sequence 5 (Experimental): Dosing Period 1 - 500 mg CK-2017357; Dosing Period 2 - Placebo; Dosing Period 3 - 375 mg CK-2017357
  Interventions: Drug: Placebo; Drug: 375 mg CK-2017357; Drug: 500 mg CK-2017357
- Treatment Sequence 6 (Experimental): Dosing Period 1 - 500 mg CK-2017357; Dosing Period 2 - 375 mg CK-2017357; Dosing Period 3 - Placebo
  Interventions: Drug: Placebo; Drug: 375 mg CK-2017357; Drug: 500 mg CK-2017357

INTERVENTIONS:
Drug: Placebo — Matching placebo in capsules administered as a single oral dose.
Drug: 375 mg CK-2017357 — 375 mg CK-2017357 in capsules administered as a single oral dose.
  Other Names: tirasemtiv
Drug: 500 mg CK-2017357 — 500 mg CK-2017357 in capsules administered as a single oral dose.
  Other Names: tirasemtiv

SUMMARY:
The primary objective of this early-stage clinical study is to demonstrate an effect of single doses of CK-2017357 on measures of skeletal muscle function and fatigability in patients with peripheral artery disease and symptomatic claudication.

DETAILED DESCRIPTION:
This study is a Phase II, double-blind, randomized, placebo-controlled, three-way crossover design of two single doses of CK-2017357 in patients with peripheral artery disease and symptomatic claudication. 36 to 72 patients will be randomized at approximately 15 study centers to one of six different treatment sequences. Each treatment sequence consists of three dosing periods in which patients receive single oral doses of placebo, 375 mg and 500 mg of CK-2017357. All six treatment sequences will enroll approximately the same number of patients. A wash out period of at least 6 days (to a maximum of 10 days) will be employed between the individual doses for each patient. This study is designed to assess the effects of CK-2017357 on measures of endurance/fatigue, work output, and walking capacity. The PK and PD relationship of CK-2017357 after two single doses will be assessed versus placebo, and the CK-2017357 concentration versus time data obtained in this study may be used to develop a population PK model to estimate intra- and inter-patient variability of PK parameters in patients with claudication.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to comprehend and willing to sign an Informed Consent Form (ICF)
2. Ability to understand written and oral English language
3. Peripheral arterial disease defined as an ankle-brachial index (ABI) at rest ≤ 0.90 in at least one leg in which the patient experiences claudication
4. Stable claudication symptoms over past 6 months (Fontaine Stage II) in at least one calf muscle due to documented peripheral artery disease
5. Females (of non-childbearing potential) or males who are 40 years of age or older
6. Body mass index (BMI) of 18.0 to 30.0 kg/m2, inclusive
7. Ability to perform the bilateral heel raise familiarization sufficient to induce typical claudication at a contraction frequency of once every other second
8. Ability to complete a six-minute walking test
9. Pre-study clinical laboratory findings (including troponin I [TnI] and creatine phosphokinase [CPK]) within the normal range, or if outside of the normal range, deemed not clinically significant by the Investigator and Sponsor's Medical Monitor
10. For female patients only: Non-childbearing potential (e.g., documented post-menopausal ≥ 1 year, sterilized, status-post hysterectomy) For male patients only: Agreement either

    * To use a condom during sexual intercourse with female partners who are of reproductive potential and to have female partners use an additional effective means of contraception (e.g., diaphragm plus spermicide, or oral contraceptives) for the duration of the study and 10 weeks after the end of the study or
    * To abstain from sexual intercourse for the duration of the study and 10 weeks after the end of the study

Exclusion Criteria:

1. Asymptomatic peripheral artery disease classified as Fontaine Stage I
2. Critical leg ischemia classified as Fontaine Stage III-IV (rest pain, tissue necrosis or gangrene)
3. Non-atherosclerotic causes of arterial occlusive disease
4. "Atypical leg pain," defined as significant residual leg discomfort at rest
5. Leg, hip, or knee surgery within 6 months prior to randomization
6. Any revascularization procedure (coronary or peripheral) within 3 months prior to randomization
7. Life-threatening ventricular arrhythmias, unstable angina, stroke, and/or myocardial infarction within 3 months prior to randomization
8. Moderate/severe symptomatic heart failure defined as NYHA Class III or IV; in patients with NYHA Class I or II heart failure, the screening heel raise familiarization must elicit claudication symptoms and not cardiac symptoms
9. Severe COPD or other respiratory impairment defined as receiving supplemental oxygen therapy at home or by clinical assessment of the Investigator
10. Poorly controlled hypertension (defined as supine resting BP >180 mmHg systolic or > 100 mmHg diastolic, or both)
11. Hypotension (defined as supine resting BP < 95 mmHg systolic or < 55 mmHg diastolic, or both, or symptomatic hypotension [standing, supine, or orthostatic])
12. Exercise tolerance (including ability to perform heel raise and six-minute walk test) that, in the opinion of the Investigator, is significantly limited by other co-morbid conditions or diseases other than claudication
13. Type 1 diabetes (juvenile onset, insulin-dependent), or poorly controlled Type 2 diabetes (defined as HbA1c > 9.0% in the past 3 months)
14. Hepatic insufficiency (defined as ALT or AST > 3x ULN, or total bilirubin > 3 mg/dL)
15. Renal insufficiency (defined as serum creatinine > 2.5 mg/dL or receiving dialysis)
16. Anemia (defined as hemoglobin < 12.0 g/dL)
17. Participation in any other investigational study drug or device trial in which receipt of an investigational study drug or device occurred within 30 days prior to dosing
18. Previous treatment with gene therapy or other vascular endothelial growth factor (VEGF)-related therapy
19. Any prior treatment with CK-2017357
20. Recent history of alcoholism or drug abuse, or significant behavioral or psychiatric problems, or other conditions which in the Investigator's opinion may impair ability to adequately comply with the requirements of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Effect of single dose of CK-2017357 on number of contractions, time and work to onset of claudication during bilateral heel raises | 1 day
  Heel raises will be monitored by an electrogoniometer placed on the index leg and performed once every other second until onset of claudication pain or fatigue as determined by electrogoniometry
Effect of single dose of CK-2017357 on number of contractions, time and work to intolerable claudication pain or maximal calf muscle fatigue | 1 day
  Heel raises will be monitored by an electrogoniometer placed on the index leg and performed once every other second until limited by intolerable claudication pain or fatigue as determined by electrogoniometry
Effect of single dose of CK-2017357 on Six-Minute Walk Test | 1 day
  Patient's self-paced walking distance over 6 minutes

SECONDARY OUTCOMES:
Characterize the relationship, if any, between the plasma concentrations of CK-2017357 and number of contractions, time and work to onset of claudication during bilateral heel raises | 1 day
  Bilateral heel raise assessments will be paired with PK concentrations obtained at or near the same time as the bilateral heel raises assessments and analyzed for concentration related effects
Characterize the relationship, if any, between the plasma concentrations of CK-2017357 and number of contractions, time and work to intolerable claudication pain or maximal calf muscle fatigue during bilateral heel raises | 1 day
  Bilateral heel raise assessments will be paired with PK concentrations obtained at or near the same time as the bilateral heel raises assessments and analyzed for concentration related effects
Characterize the relationship, if any, between the plasma concentrations of CK-2017357 and Six-Minute Walk Test | 1 day
  Six-Minute Walk Test will be paired with PK concentrations obtained at or near the same time Six Minute Walk Test and analyzed for concentration related effects
Number of patients with adverse events | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Hiatt, MD, Study Director — Colorado Prevention Center; Alan Hirsch, MD, Principal Investigator — University of Minnesota
Locations (14):
- United States (14):
  - Tatum Ridge Internal Medicine, Phoenix, Arizona
  - Apex Research Institute, Santa Ana, California
  - Stanford Hospital and Clinics, Stanford, California
  - Denver Health Medical Center, Denver, Colorado
  - Tampa Bay Medical Research, Clearwater, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - DMI Research, Inc, Pinellas Park, Florida
  - Maine Research Associates, Auburn, Maine
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Baylor College of Medicine, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - National Clinical Research - Norfolk, Inc., Norfolk, Virginia
  - National Clinical Research - Richmond, Inc., Richmond, Virginia

REFERENCES:
- [Result] Hiatt WR, Hirsch AT, Bauer TA, Malik F, Lee J, Lin Y, Han FX, Chen MM, Jones D, Cedarbaum JM, Wolff AA. Efficacy and Tolerability of the Novel Fast Skeletal Muscle Troponin Activator, CK-2017357, in Patients with Claudication. 22nd Annual Sessions of the Society for Vascular Medicine. Boston, MA, June 2011
- [Derived] Bauer TA, Wolff AA, Hirsch AT, Meng LL, Rogers K, Malik FI, Hiatt WR. Effect of tirasemtiv, a selective activator of the fast skeletal muscle troponin complex, in patients with peripheral artery disease. Vasc Med. 2014 Aug;19(4):297-306. doi: 10.1177/1358863X14534516. Epub 2014 May 28. PMID 24872402